CLINICAL TRIAL: NCT05455580
Title: Nurses Taking On Readiness Measures - Mercer County, New Jersey
Acronym: NTORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Tara Heagele, Assistant Professor, Hunter College of City University of New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0097
Record Dates: First submitted 2022-06-09; First posted 2022-07-13 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Disaster; Vulnerable Populations
Keywords: disabled persons; civil defense; hazard; emergency; preparedness; planning; readiness; kit; disaster planning; emergency preparedness
MeSH Terms: conditions — Emergencies; Piebaldism

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, non-blinded, quasi-experimental, pre- and post-test phase I feasibility design pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-TORM Intervention (Experimental): This is a non-randomized, non-blinded, quasi-experimental, pre- and post-test phase I feasibility design pilot study.
  Interventions: Behavioral: Nurses Taking On Readiness Measures (N-TORM)

INTERVENTIONS:
Behavioral: Nurses Taking On Readiness Measures (N-TORM) — The intervention will begin with instructing the participant to complete the Family Disaster Plan booklet. The principal investigator will talk about the different sections of the booklet and instruct the participants how to fill out their emergency plans. Participants will write their medical history, medications, physician, next of kin, pharmacy contact information, evacuation plan information, family communication plan, and insurance policy numbers and contact information. The booklet includes household emergency preparedness recommendations, evacuation zone information, a disaster supply kit contents list, local utility company contact information, shelter locations, and special needs and priority utility restoration registry information. The participants will be provided with a disaster supply kit after successful completion of the booklet. The disaster supply kit is part of the intervention and is not considered compensation.

SUMMARY:
Nurses Taking On Readiness Measures (N-TORM) is an innovative nurse-driven household emergency preparedness (HEP) intervention modeled after an existing community intervention provided by emergency management personnel. This phase I feasibility pilot study will describe the implementation and effectiveness of N-TORM in the community setting, but provided by nurses. The aims of this implementation study are to: (a) increase the reach of N-TORM to vulnerable populations; (b) evaluate the effectiveness of N-TORM for increasing HEP knowledge and behavior; (c) implement N-TORM in a community located in an area at increased risk for disasters, measuring consistency of delivery, time, and cost of N-TORM; (d) describe the factors necessary to maintain and expand N-TORM, and; (e) pilot test a new HEP instrument in order to perform psychometric testing on the instrument and generate reliability and validity data.

DETAILED DESCRIPTION:
As more chronically ill people are living in the community and disasters are occurring frequently, the elderly and the medically frail vulnerable populations are experiencing significantly more disaster-related morbidity and mortality than the rest of the population. Lack of knowledge on how best to prepare for disasters and lack of means to purchase supplies are significant barriers to adequate household emergency preparedness (HEP). Community-based HEP interventions present a unique opportunity to address these barriers and disaster-related morbidity and mortality disparities in vulnerable populations. Modeled after a community intervention targeting healthy seniors (Golden, 2013) and residents (New York State, n.d.), Nurses Taking On Readiness Measures (N-TORM) is a nurse-driven HEP intervention that will be offered in the community to older adults, individuals with chronic illnesses, pregnant women, and caregivers of medically frail individuals. The Federal Emergency Management Agency (FEMA) Emergency Management Institute (2014) states that these individuals have access or functional needs during disasters and are considered vulnerable populations. The proposed study develops, tests, and evaluates the N-TORM intervention for the purpose of contributing to generalizable knowledge about the nurses' role in the HEP of vulnerable community members. The proposed phase I feasibility pilot study will specifically target independently living community members with access and functional needs. The N-TORM intervention will enable the household to meet the FEMA recommendations for HEP, to safely shelter in place, and evacuate quickly with their supplies if needed. Measurable outcomes of the proposed study include the nurse's impact on the participants' level of HEP post-intervention and participant satisfaction with the intervention. Multi-disciplinary collaboration with engagement of community and government organizations will be demonstrated by the proposed study. Community resources provided by the New Jersey Office of Emergency Management will be incorporated into N-TORM. It is plausible that the long-term impact of the N-TORM intervention would be lives saved and resources conserved. Because the N-TORM intervention uses an all-hazards approach, it is possible to replicate nationally and with different vulnerable populations.

* RQ 1: What is the baseline level of HEP of the participants?
* RQ 2: How much of the variance in HEP is explained by the Household Emergency Preparedness Instrument (HEPI)?
* RQ 3: Is there a significant difference in HEP level after receiving the N-TORM intervention?
* RQ 4: What are the facilitators and barriers of nurses delivering and participants receiving the N-TORM intervention? Finally, the proposed study will also pilot test a new household emergency preparedness instrument (Heagele et al., 2020) in order to perform psychometric testing on the instrument and generate reliability and validity data.

Potential Participants will be recruited from a private Facebook group called "Hamilton Twp. Mercer County NJ." The principal investigator will also utilize the Snowball Sampling technique where participants suggest other potential participants. The principal investigator will provide flyers to the participants with the hope that they will share them with other potential participants.

The principal investigator will then perform the online screening. The principal investigator will deliver the recruitment script to eligible participants.

Participants will be consented only once when they enroll in the study. The consent form will be provided during the online screening/recruitment for the potential participant to read. The consent form will be signed at the in-person meeting at a public place of the participant's choice within Mercer County, New Jersey, after the principal investigator has answered any questions that the participant has.

After informed consent is obtained, the principal investigator will perform the study procedures with the participant:

1. administer the demographic data form to the participants.
2. administer the Household Emergency Preparedness Instrument (HEPI) to the participants before and after the intervention.
3. perform the N-TORM intervention.
4. administer the participant experience survey. The completed Family Disaster Plan booklets will not be copied, collected, stored, or used for research purposes. The booklets are for the participants to keep; they are the participants' household emergency preparedness plans and they will also serve as a community disaster resources information source. The participants will be provided with a disaster supply kit after successful completion of the booklet. The disaster supply kit, valued at $111.60 on September 18, 2020, is part of the intervention and is not considered compensation.

There is no need for follow-up with the participants after they have completed the intervention.

There is no more than minimal risk for participation in this study. Little to no feelings of discomfort are expected. When completing the HEPI and the Family Disaster Plan booklet, participants may experience unpleasant memories, anxiety, or respondent burden. To mitigate this risk, participants will be able to skip HEPI questions or stop the HEPI at any time if they become uncomfortable. Participants will also be able to stop filling out the Family Disaster Plan booklet at any time. In addition, the informed consent includes an assurance of the participant's right to choose not to participate or to terminate participation at any time during the intervention and states that, should the participant decide not to participate in this research study, his or her relationship with the study team will not change and he or she will not lose any benefits to which he or she is otherwise entitled.

There are no direct benefits to participating in this study. This research does not claim to present a therapeutic benefit to the participants. Participants who successfully complete the intervention may be self-sufficient for up to 72-hours post-disaster, but the association between disaster preparedness level and disaster resilience has not been empirically tested. It is anticipated that this study will benefit society. The study data can build evidence for a promising individual and community HEP intervention. This HEP intervention can also be used in longitudinal studies to determine whether there is an association between being prepared for a disaster and surviving the disaster without the need for rescue or outside assistance. For medically frail community members, it can be determined whether there is an association between being prepared for a disaster and surviving the disaster without an acute exacerbation of a chronic illness and with no change in baseline functional status.

The participants will not incur any research-related costs. The participants will not be compensated for their participation.

The data from the HEPIs, demographic data forms, and surveys will be transcribed by the principal investigator into electronic documents. This deidentified data will be stored on a password-protected, encrypted server, which complies with the City University of New York's Computer Use and Internet-Based Research Policy, for three years after the study is completed and closed out with the IRB. After the three years are completed, the study data will be deleted. The paper copies of the HEPIs, demographic data forms, and surveys will be shredded after they are transcribed. The data will not be stored or distributed for future research studies.

The investigators will analyze the quantitative and qualitative data. A statistician will be utilized to assist with analyzing deidentified quantitative data. The reliability of the HEPI will be measured by looking at the internal consistency of the items. Polychoric correlations will be used to examine the factor structure of the HEPI. Known-group validity of the HEPI will be assessed by comparing the scores of the participants who self-reported that they were unprepared for a disaster before and after the N-TORM intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* have access and functional needs during disasters or are caregivers of individuals with access and functional needs
* live independently within Mercer County, New Jersey (i.e., not in a rehabilitation facility, long-term care facility, halfway house, or prison)
* consent to participate

Exclusion Criteria:

* cognitive impairments
* less than 18 years of age
* Non-English speaking
* Non-English reading families

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara N Heagele, PhD, Principal Investigator — City University of New York, School of Public Health
Locations (1):
- Hunter College, City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golden, S. (2013). STORM Seniors Taking on Readiness Measures: Family disaster plan. Freehold, NJ Monmouth County Sheriff's Office.
- [Background] Heagele TN, McNeill CC, Adams LM, Alfred DM. Household Emergency Preparedness Instrument Development: A Delphi Study. Disaster Med Public Health Prep. 2022 Apr;16(2):570-582. doi: 10.1017/dmp.2020.292. Epub 2020 Nov 20. PMID 33213596
- [Background] Heagele TN, Nurse-Clarke NJ. A Nurse-Led Home Disaster Preparedness Intervention for New Parents. Neonatal Netw. 2022 Jan 1;41(1):5-10. doi: 10.1891/11-T-714. PMID 35105790
- [Background] Heagele TN, Adams LM, McNeill CC, Alfred DM. Validation and Revision of the Household Emergency Preparedness Instrument (HEPI) by a Pilot Study in the City University of New York. Disaster Med Public Health Prep. 2022 Mar 25;17:e126. doi: 10.1017/dmp.2022.35. PMID 35332858
- See also: New York State Citizen Preparedness Corps. — https://www.dhses.ny.gov/citizen-preparedness-corps
- See also: FEMA Emergency Management Institute. (2014). IS-368: Including people with disabilities and others with access and functional needs in disaster operations. — https://training.fema.gov/is/courseoverview.aspx?code=is-368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and data collection began in March 2022 and concluded in May 2022. We recruited potential participants from a private Facebook group created for local residents to discuss concerns and share events happening in the county. Because we experienced difficulty with finding participants willing to travel to meet an unfamiliar interventionist from a social media post, we also utilized snowball sampling.
Pre-assignment Details: Participants with cognitive impairments were excluded because they are not responsible for their preparedness activities. However, their primary caregivers were eligible to participate.
Period: Overall Study
Arm/Group | N-TORM Intervention
Started | 31 (March 2022)
Completed | 31 (Recruitment ceased in May of 2022 at 31 successful completions of the N-TORM intervention, which was the number of disaster kits procured for this feasibility study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Mean age of the respondents was 51 years, and they reported having lived an average of 12 years in their current home and 18 years in their current community. The majority identified as female (n = 24, 77%), white (n = 27, 87%), and that they spoke English as their first language (n = 28, 90%). Most (n = 17, 55%) were married.
Arm/Group | N-TORM Intervention
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Native | 1
  Asian | 1
  Black | 2
  Latin | 2
  White | 27
Years in home [Mean (Standard Deviation); unit: years] — Years lived in the home (continuous)
  years | 12.3 (14.2)
Years in community [Mean (Standard Deviation); unit: years] — Years lived in the community (continuous)
  years | 18.1 (17.2)
Relationship [Count of Participants; unit: Participants]
  Married | 17
  Widowed | 1
  Divorced | 5
  Domestic partner or civil union | 1
  Single with significant other | 3
  Single, never married | 4
Employment [Count of Participants; unit: Participants]
  Full-time | 21
  Not employed | 3
  Retired | 6
  Disabled | 1
Education [Count of Participants; unit: Participants]
  High school diploma or GED | 3
  Some college | 4
  Associate degree | 2
  Baccalaureate degree | 14
  Graduate degree | 8
Income [Count of Participants; unit: Participants]
  < $20,000 | 2
  $20-34,999 | 1
  $35-49,999 | 1
  $50-74,999 | 7
  $75-99,999 | 6
  $100-149,999 | 9
  $150,000 or more | 5
Home ownership [Count of Participants; unit: Participants]
  Own | 22
  Rent | 8
  Other | 1
Structure [Count of Participants; unit: Participants] — Type of home
  Participants
    Detached single | 21
    Multi, 1-2 stories | 7
    Multi, 3 or more stories | 1
    Mobile or manufactured | 1
    No response | 1
Uses medications [Count of Participants; unit: Participants] — Dependent on at least one prescription medication
  Participants
    Yes | 30
    No | 1
Uses medical equipment [Count of Participants; unit: Participants]
  Yes | 12
  No | 19
Has a disability [Count of Participants; unit: Participants]
  Yes | 4
  No | 27
Served in the military [Count of Participants; unit: Participants]
  Yes | 2
  No | 29
First language is English [Count of Participants; unit: Participants]
  Yes | 28
  No | 3

OUTCOME MEASURES:

1. Primary Outcome: Household Emergency Preparedness Instrument (HEPI) Score
Description: The Household Emergency Preparedness Instrument (HEPI) is an all-hazards, comprehensive, 51-question instrument used to ascertain if a respondent is prepared for disasters. Higher scores on the HEPI indicate higher levels of preparedness. Excluding the Access and Functional Needs (AFN) and Special Actions (SA) subscales that are not applicable to all respondents, the minimum score a participant could receive on the General Preparedness (GP) scale is 0 and the maximum score is 40 (1 point for each yes-response and 0 points for each no-response). There is support for face, content, and criterion validity of this instrument. The HEPI questions are objective and ask about what the respondent presently owns or does in a dichotomous format.
Time Frame: Baseline (Pre-test) and approximately 30 minutes (Post-test)
Population: Inclusion criteria for the participants was being aged 18 years or older, English-speaking, medically frail (i.e., having access and functional needs during disasters) or were caregivers of individuals with access and functional needs, living independently (i.e., not in a rehabilitation facility, long-term care facility, halfway house, or prison) within one county in New Jersey, and self- identifying as feeling unprepared for disasters.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-TORM Intervention
Number analyzed (Participants) | 31
score on a scale
  Pre-test - HEPI General Preparedness Scale | 5.5 (4.1)
  Post-test - HEPI General Preparedness Scale | 20.2 (3.1)

ADVERSE EVENTS:
Time Frame: During 30-minute intervention
Description: No adverse events occurred.
Arm/Group | N-TORM Intervention
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT05455580/Prot_SAP_ICF_000.pdf